CLINICAL TRIAL: NCT03889223
Title: Ultrasonographic and Comfort Comparison of Sitting Fetal Cross-legged Position With Lateral Decubitus Fetal Position on Healthy Volunteers; a Randomized, Consecutive-controlled Clinical Trial
Brief Title: Ultrasonographic and Comfort Comparison of Sitting Fetal Cross-legged Position With Lateral Decubitus Fetal Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Fatma Ferda Kartufan, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: KAEK- tez
Record Dates: First submitted 2019-03-12; First posted 2019-03-26 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia, Conduction
Keywords: neuraxial anesthesia positioning technique; sitting cross-legged fetal position; lateral decubitus fetal position; ultrasonography

STUDY DESIGN:
Intervention Model Description: Systematic randomization was made from 150 volunteers, and 50 participants were chosen. All 50 participants were planned to sit on the stretcher in both of the two positioning techniques sequentially (one after another). The two positioning techniques are SCF and LDF. The investigator was planned to record all of the participants' anatomical measurements in both of those positioning techniques evaluated via ultrasonography. After each position participants were planned to evaluate each positioning technique's comfort by 7-point numerical rating scale from minimum
  1 meaning "very bad" to maximum 7 meaning "excellent."
Who Masked: Outcomes Assessor
Masking Description: The ultrasonography was made by a consultant radiologist (M.D.) The consultant didn't know which position was for control and which was the one the study evaluates. Although investigators were trying to mask the outcomes assessor; the consultant saw the positions because there is no way to hide the sitting positions of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The LDF neuraxial positioning technique (Active Comparator): In the LDF neuraxial positioning technique, fifty participants were planned to lay down the stretcher facing the wall of the sonography room and turned back to the consultant Radiologist. Volunteers jaw touch to chest and legs in abdominal flexion with hands are on the knees. The position is completed with the back curved in the fetal position. Then the USG is performed by the consultant Radiology M.D. in maximum 2 hours time to each participant, and the 7-point NRS evaluation is done by each participant in maximum 30 minutes time until the study ends within 15 weeks.
  Interventions: Procedure: Anatomical intervention with USG and comfort evaluation with NRS
- The SCF neuraxial positioning technique (Experimental): In the SCF neuraxial positioning technique, the same fifty participants were planned to sit on the same part of the stretcher facing the wall of the sonography room and turned back to the consultant Radiologist with legs crossed, forearms of the participants are on the lap and hands are on the knees, and the position is completed with the back curved in the fetal position.Then the USG is performed by the consultant Radiology M.D. in maximum 2 hours time to each participant, and the 7-point NRS evaluation is done by each participant in maximum 30 minutes time until the study ends within 15 weeks.
  Interventions: Procedure: Anatomical intervention with USG and comfort evaluation with NRS

INTERVENTIONS:
Procedure: Anatomical intervention with USG and comfort evaluation with NRS — The anatomical evaluation of the two neuraxial positioning techniques sonographically and comparison of comfort with the 7-point NRS

SUMMARY:
A prosperous neuraxial anesthesia positioning ensures a raised chance of successful needle placement. The primary aim is to compare "Sitting Cross-legged Fetal Position -SCF" with "Lateral Decubitus Fetal Position-LDF" anatomically via sonography.

Secondary aim is to compare their comfort.

DETAILED DESCRIPTION:
Fifty participants were included to this prospective, randomized, consecutive controlled clinical study. Six parameters were evaluated in each position; subcutaneous tissue (ST), skin to spinous process (S-SP), transverse diameters of bilateral paraspinal muscles (left paraspinal muscle [LPM] and right paraspinal muscle [RPM]), interspinous gap opening (ISGO), mean of bilateral paraspinal muscles (MPM). The change of every measurement recorded via ultrasonography (USG) according to the positioning techniques were also calculated. The calculations are explained briefly in primary outcomes (including the change of SCF-LDF in ST, S-SP, LPM, RPM, MPM, ISGO). Stretcher comfort (SC), position comfort (PC), lumbar comfort (LC), and abdominal comfort (AC) were evaluated by the participants with the 7-point Numerical Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* healthy and adult volunteers,
* must be able to do the sitting cross-legged fetal position ( SCF ),
* must be able to do the Lateral decubitus fetal position (LDF).

Exclusion Criteria:

* Lumbar hernia,
* Scoliosis,
* History of spine surgery,
* History of trauma,
* History of lower back pain,
* Arthropathy {especially pelvic or knee problems},
* Could not be able to do one or both of the two neuraxial position techniques.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Interspinous gap opening (ISGO) measurement in the SCF | For the SCF technique, ISGO is measured in the first 10 minutes(mins.) time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the wideness measurement of the ISGO in millimeters via ultrasonography (USG) in the SCF
Left paraspinal muscle (LPM) measurements in the SCF | For the SCF technique, LPM is measured between the 10th and 20th mins. of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the diameter measurement of the LPM in millimeters via ultrasonography in the SCF
Right paraspinal muscle (RPM) measurements in the SCF | For the SCF technique, RPM is measured in between the 20th and 30th mins. of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the diameter measurement of the RPM in millimeters via ultrasonography in the SCF
The mean of bilateral paraspinal muscles (MPM) in the SCF | For the SCF technique, MPM measurement is planned to be done in between the 30th and 40th mins. of the study,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by ( [LPM+RPM]/2) in millimeters in the SCF
Subcutaneous tissue (ST) measurements in the SCF | For the SCF technique, ST measurement is planned to be done in between the 40th and 50th mins. of the study,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the thickness measurement of the subcutaneous tissue in millimeters via ultrasonography in the SCF
The skin to spinous process (S-SP) measurements in the SCF | : For the SCF technique, S-SP measurement is planned to be done in between the 50th and 60th mins. of the study,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the depth measurement of the skin to spinous process in millimeters via ultrasonography in the SCF
Interspinous gap opening (ISGO) measurement in the LDF | ISGO measurement in the LDF will be done right after NRS evaluation of the SCF, in between the 70th and 80th mins. of the study,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the wideness measurement of the ISGO in millimeters via ultrasonography in the LDF
Left paraspinal muscle (LPM) measurements in the LDF | LPM measurement in the LDF will be done in between the 80th and 90th mins. of the study,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the diameter measurement of the LPM in millimeters via ultrasonography in the LDF
Right paraspinal muscle (RPM) measurements in the LDF | RPM measurement in the LDF will done in between the 90th and 100th mins. of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant through study completion up to 20 weeks.
  the diameter measurement of the RPM in millimeters via ultrasonography in the LDF
The mean of bilateral paraspinal muscles (MPM) in the LDF | MPM measurement in the LDF will be done in between the 100th and 110th mins. time of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by ( [LPM+RPM]/2) in millimeters in the LDF
Subcutaneous tissue (ST) measurements in the LDF | ST measurement in the LDF will be done in between the 110th and 120th mins. time, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the thickness measurement of the subcutaneous tissue in millimeters via ultrasonography in the LDF
The skin to spinous process (S-SP) measurements in the LDF | S-SP measurement in the LDF will be done in between the 120th and 130th mins. of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  the depth measurement of the skin to spinous process in millimeters via ultrasonography in the LDF
the change of ISGO (ISGO SCF-LDF) | ISGO in the SCF measured in the first 10mins., and ISGO in the LDF measured in between the 70th and 80th mins. of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation; ([ISGO in the SCF in millimeters]-[ISGO in the LDF in millimeters])
the change of LPM (LPM SCF-LDF ) | LPM in the SCF measured in between the 10th and 20th mins., and LPM in the LDF measured in between the 80th and 90th mins., in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation; ([LPM in SCF in millimeters]-[LPM in LDF in millimeters])
the change of RPM (RPM SCF-LDF) | RPM in the SCF measured in between the 20th and 30th mins., and RPM in the LDF measured in between 90th and 100th mins., in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation ([RPM in SCF in millimeters]-[RPM in LDF in millimeters])
the change of MPM (MPM SCF-LDF) | MPM in the SCF measured in between the 30th and 40th mins., and MPM in the LDF measured in between 100th and 110th mins., in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation ([MPM in SCFin millimeters]-[MPM in LDF in millimeters])
the change of ST (ST SCF-LDF) | ST in the SCF measured in between the 40th and 50th mins., and ST in the LDF measured in between the 110th and 120th, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation ([ST in SCF in millimeters]-[ST in LDF in millimeters])
the change of S-SP (S-SP SCF-LDF) | S-SP in the SCF measured in between the 50th and 60th mins., and S-SP in the LDF measured in between the 120th and 130th mins., in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Measured by calculation ([S-SP in SCF in millimeters]-[S-SP in LDF in millimeters])

SECONDARY OUTCOMES:
Comfort evaluation in the SCF via 7-point numerical rating scale (NRS) | NRS measurement is planned to be done right after the SCF position in between the 60th and 70th mins. time,in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks..
  Comfort evaluation of the SCF technique is planned to be done by the participant right after USG. The 7-point NRS includes 7 scale. The minimum scale is"1" means very bad, "2" means bad, "3" means fair, "4" means normal, "5" means good, "6" means very good, and the maximum scale is "7" means excellent.
Comfort evaluation in the LDF via 7-point numerical rating scale (NRS) | NRS measurement is planned to be done right after the LDF position in between the 130th and 140th mins. time of the study, in 10 mins. time of the total 3hr and 30 mins. study, for each participant, through study completion up to 20 weeks.
  Comfort evaluation of the LDF technique is planned to be done by the participant right after USG. The 7-point NRS includes 7 scale. The minimum scale is"1" means very bad, "2" means bad, "3" means fair, "4" means normal, "5" means good, "6" means very good, and the maximum scale is "7" means excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Ferda Kartufan, Assist.Prof., Principal Investigator — Anesthesiology and Reanimation Department; Feyza Aksu, MD, Study Chair — Anesthesiology and Reanimation Department; Özge Köner, Prof., Study Director — Anesthesiology and Reanimation Department; Ayşegül Görmez, Consult.MD, Study Chair — Radiology Department
Locations (1):
- Yeditepe University Hospital, Istanbul, İçerenköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dimaculangan DP, Mazer JA, Maracaja-Neto LF. Sonographic evaluation of lumbar interlaminar space opening in a variety of patient body positions for optimal neuraxial anesthesia delivery. J Clin Anesth. 2016 Nov;34:159-65. doi: 10.1016/j.jclinane.2016.03.045. Epub 2016 May 6. PMID 27687365